CLINICAL TRIAL: NCT04473521
Title: A Clinical Study Assessing Maximum Maxillary Bite Force When Using a Novel Denture Adhesive Compared to Using No-adhesive
Brief Title: A Clinical Study to Assess Force Required to Dislodge Upper Denture With and Without Use of a Novel Denture Adhesive
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study objectives no longer met business need
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 213629
Record Dates: First submitted 2020-06-29; First posted 2020-07-16 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Denture Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Adhesive (No Intervention): No adhesive will be applied.
- Super Poligrip Free (SPF) (Active Comparator): The denture adhesive of 1.00grams (g) +/- 0.05g will be applied to only the maxillary denture in long, continuous strips manner that is controlled by weight for the maxillary dentures. Mandibular denture will be stabilised using this adhesive up to 2 times (maximum [max] 3 adhesive applications per day) at examiner's discretion.
  Interventions: Device: Super Poligrip Free
- Investigational Adhesive (Experimental): The denture adhesive of 1.00g +/- 0.05g will be applied only to the maxillary denture only in long, continuous strips manner that is controlled by weight for the maxillary dentures. Mandibular denture will be stabilized using SPF adhesive up to 2 times (max 3 adhesive applications per day) at examiner's discretion.
  Interventions: Device: Investigational denture adhesive cream
- Investigational Adhesive + Hot drink (Experimental): The denture adhesive of 1.00g +/- 0.05g will be applied to only the maxillary denture in long, continuous strips manner that is controlled by weight for the maxillary dentures. Hot drinks will be provided within 1 hour of completing lunch and dinner and must be consumed within 30 minutes. Mandibular denture will be stabilized using SPF adhesive up to 2 times (max 3 adhesive applications per day) at examiner's discretion.
  Interventions: Device: Investigational denture adhesive cream

INTERVENTIONS:
Device: Investigational denture adhesive cream — The denture adhesive application will be controlled by weight (1.00g +/-0.05g) applied to the maxillary denture only.
  Arms: Investigational Adhesive; Investigational Adhesive + Hot drink
Device: Super Poligrip Free — The denture adhesive application will be controlled by weight (1.00g +/- 0.05g) applied to the maxillary denture only.
  Arms: Super Poligrip Free (SPF)

SUMMARY:
The purpose of this study is to investigate the hold properties of an investigational denture adhesive using an established methodology called the maximum incisal bite force (BF), and Kapur-Olshan (KO) index for denture retention and stability. The effects of hot drinks and two questionnaires relating to participants' perception will also be assessed for the investigational denture adhesive.

DETAILED DESCRIPTION:
This study will be a single-centre, controlled, randomized, single blind, 4-treatment, 4-period, cross-over study to evaluate maximum maxillary bite force in a population of full maxillary denture wearers. This study consists of 5 visits (1 screening visit and 4 treatment periods including minimum washout period of 2 days between treatment visits). Participant's maxillary and mandibular dentures will be assessed for retention and stability using KO index and whether they are well made. Participants will be randomized to one of the 4 treatment groups i.e. No adhesive, Super Poligrip Free (SPF), Investigational Adhesive and Investigational Adhesive + Hot drink arm group and will undergo an oral soft tissue (OST) and Oral Hard Tissue (OHT) examination. Participants who will meet all the inclusion and no exclusion criteria will continue the study. Participants will complete the BF measurement, KO assessment, OST, OHT examination and participants 'perception questionnaire as per the schedule.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant with a completely edentulous maxillary arch restored with a conventional maxillary full denture with an acrylic base. The maxillary denture prosthesis must fulfil all of the following:

  1. At least moderately well-fitting (Kapur Index, Olshan Modification: retention score greater than or equal to (>=)2, stability score >=2) at the Screening (V1) visit,
  2. Are well made (according to the well-made assessment).
* Participant with BF measurements which satisfy the following criteria:

  1. The "qualifying" BF measurements (without adhesive) at V1 must be less than or equal to (=<)9lbs.
  2. At least 2 of the 4 "qualifying" BF measurements (without adhesive) at V1 (Screening) must be reproducible (within +/-2lbs).
  3. The "Baseline" BF measurement (without adhesive) at V2-5 must be <=9lbs.
  4. The "Baseline" BF measurement (without adhesive) at V2-5 and at least 1 of the 3 "practice" BF measurements must be within +/-2lbs of each other.
* A participant who is dentate in the mandibular arch or has a partial or full denture in the mandibular arch that is:

  1. sufficiently stable, in the opinion of the investigator, to enable the bite force determination to be performed.
  2. well made (according to the well-made assessment).

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* A participant who is currently taking or has taken a bisphosphonate drug (i.e., Fosamax, Actonel, Boniva).
* Use of any medication or condition (e.g. insulin dependent diabetes) that, in the opinion of the investigator, would interfere with the conduct of the study.
* A participant who has any clinically significant or relevant oral abnormality (e.g. temporomandibular joint [TMJ] problems) that, in the opinion of the investigator, could affect the participant's participation in the study.
* A participant clinically identified as having an incisal bite relation or any other tooth abnormality which could affect the BF measurements or participant safety.
* A participant who has any condition or medication which, in the opinion of the investigator, is currently causing xerostomia or which would interfere with the conduct of the study.
* A participant with a recent history (within the last year) of alcohol or other substance abuse.
* A participant with OST examination findings (at V1) such as stomatitis, open sores, lesions, cavitied caries lesions, redness or swelling which in the opinion of the investigator, would interfere with the conduct of the study.
* A participant who has previously been enrolled in this study.
* Any participant who can't comply with study requirements and/or who would not be able to reliably perform a valid bite at the examiner's discretion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-04 (Estimated); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
Area Over Baseline Over 12 Hours (AOB 0-12) to Compare Maximum Incisal Bite Force (BF) | Up to 12 hours
  Incisal bite force measurements will be performed to analyse the denture dislodgement as measure of denture adhesive hold efficacy. All BF measurements will be conducted by an examiner. AOB0-12 will be used to assess the incisal bf and is defined as (AUC0-12)/12 minus baseline BF(pounds [lbs]). Area under the Curve (AUC) is calculated from 0 to 12 hours (hr) using the trapezoid method; denoted as AUC0-12. This transformation will return the measurement to the same scale as the original observations. Area over baseline in BF as measured by AOB0-12 will be analyzed for each of the three interventional products, compared to no adhesive. Higher values of AOB0-12 demonstrate a stronger bite force overtime than lower values.

SECONDARY OUTCOMES:
Area Over Baseline (AOB) at 0.5, 1, 3, 6 And 9 Hours to Compare Maximum Incisal Bite Force | Baseline, at 0.5, 1, 3, 6 and 9 hours
  Incisal bite force measurements will be performed to analyse the denture dislodgement as measure of denture adhesive hold efficacy. All BF measurements will be conducted by an examiner. This transformation will return the measurement to the same scale as the original observations. AOB for 0.5, 1, 3, 6 and 9 hours will be analyzed using the trapezoid method. Area over baseline in BF as measured by AOB will be analyzed for each of the three active products, compared to no adhesive. Higher values of AOB demonstrate a stronger bite force overtime than lower values.
Kapur Olshan (KO) Index Scores for Denture Retention | Baseline, at 3 hours
  KO Index score will be assessed to examine retention and stability performance of maxillary dentures. Retention will be measured on score of 0-5 to assess nature of resistance offered by denture to vertical force at the canine/lateral incisor region of the denture: 0= No retention- when the denture was seated in place, it displaced itself; 1= Poor- denture offers slight resistance to vertical pull and little or no resistance to lateral force; 2= Fair- denture offered moderate resistance to vertical pull and little or no resistance to lateral forces; 3= Good- denture offered moderate resistance to vertical pull and lateral force; 4= Very Good- denture offered very good resistance to vertical pull and lateral force; 5=Excellent - denture offered excellent resistance to vertical pull and lateral force. Higher the score, higher the retention ability of denture.
Kapur Olshan (KO) Index Scores for Denture Stability | Baseline, at 3 hours
  KO Index score will be assessed to examine retention and stability performance of maxillary dentures. Stability will be measured on score of 0-4: 0= No stability- when denture base had extreme rocking under pressure; 1= Poor- when denture base had moderate rocking on its supporting structures under pressure; 2= Fair- when denture base had slight rocking on its supporting structures under pressure; 3= Good- when denture base had very slight rocking on its supporting structures under pressure; 4= Excellent- when denture base offered no rocking on its supporting structures under pressure. Higher the score, higher the denture stability.
Composite Kapur Olshan (KO) Index Scores for Denture Retention and Stability | Baseline, at 3 hours
  KO Index score will be assessed to examine retention and stability performance of maxillary dentures. Retention will be measured on score of 0-5 to assess nature of resistance offered by denture to vertical force at the canine/lateral incisor region of the denture: 0=No retention; 1= Poor; 2=Fair; 3=Good; 4=Very Good;5=Excellent. Stability will be measured as score of 0-4 to assess nature of rocking offered by maxillary denture by placing alternate horizontal force at the cuspid and contralateral molar regions of the upper denture: 0=No stability; 1=Poor; 2=Fair; 3=Good; 4=Excellent. Composite KO Index scores will be measured as the sum score of retention & stability of dentures such that a sum score of zero (0) represents no retention and stability and a sum score of 9 represents excellent retention and stability.
Area Over Baseline (AOB) at 0.5, 1, 3, 6, 9 and 12 Hours to Compare Maximum Incisal Bite Force Following the Consumption of a Hot Drink | Baseline, at 0.5, 1, 3, 6, 9 and 12 hours
  Incisal bite force measurements will be performed to analyse the denture dislodgement as measure of denture adhesive hold efficacy. All BF measurements will be conducted by an examiner. This transformation will return the measurement to the same scale as the original observations. AOB for 0.5, 1, 3, 6, 9 and 12 hours will be analyzed using the trapezoid method. Change from baseline in BF as measured by AOB will be analyzed for each of the three active products, compared to no adhesive. Assessment of maximum incisal bite force of an investigational denture adhesive following the consumption of a hot drink to no adhesive was done. Higher values of AOB demonstrate a stronger bite force overtime than lower values.
Kapur Olshan (KO) Index Scores for Denture Retention Following the Consumption of a Hot Drink | Baseline, at 3 hours
  KO Index score will be assessed to examine retention and stability performance of maxillary dentures following the consumption of a hot drink versus no adhesive. Retention will be measured on score of 0-5 to assess nature of resistance offered by denture to vertical force at the canine/lateral incisor region of the denture: 0= No retention- when the denture was seated in place, it displaced itself; 1= Poor- denture offers slight resistance to vertical pull and little or no resistance to lateral force; 2= Fair- denture offered moderate resistance to vertical pull and little or no resistance to lateral forces; 3= Good- denture offered moderate resistance to vertical pull and lateral force; 4= Very Good- denture offered very good resistance to vertical pull and lateral force; 5=Excellent - denture offered excellent resistance to vertical pull and lateral force. Higher the score, higher the retention ability of denture.
Kapur Olshan (KO) Index Scores for Denture Stability Following the Consumption of a Hot Drink | Baseline, at 3 hours
  KO Index score will be assessed to examine retention and stability performance of maxillary dentures following the consumption of a hot drink versus no adhesive. Stability will be measured on score of 0-4: 0= No stability- when denture base had extreme rocking under pressure; 1= Poor- when denture base had moderate rocking on its supporting structures under pressure; 2= Fair- when denture base had slight rocking on its supporting structures under pressure; 3= Good- when denture base had very slight rocking on its supporting structures under pressure; 4= Excellent- when denture base offered no rocking on its supporting structures under pressure. Higher the score, higher the stability of denture.
Composite Kapur Olshan (KO) Index Scores for Denture Retention and Stability Following the Consumption of a Hot Drink | Baseline, at 3 hours
  KO Index score will be assessed to examine retention and stability performance of maxillary dentures following the consumption of a hot drink versus no adhesive. Retention will be measured as score of 0-5 to assess nature of resistance offered by denture to vertical force at the canine/lateral incisor region of the denture: 0=No retention; 1= Poor; 2=Fair; 3=Good; 4=Very Good;5=Excellent. Stability will be measured as score of 0-4 to assess nature of rocking offered by maxillary denture by placing alternate horizontal force at the cuspid and contralateral molar regions of the upper denture: 0=No stability; 1=Poor; 2=Fair; 3=Good; 4=Excellent. Composite KO Index scores will be measured as the sum score of retention & stability of dentures such that a sum score of zero represents no retention and stability and a sum score of 9 represents excellent retention and stability.
Number of Participants who Feel Their Denture is More Stable and Secure After Using Adhesive | Baseline, 9 hr after the BF measurement
  Denture stability and retention questionnaire will be completed by participants post dinner and hot drink after 9hr BF measurement for investigational adhesive + hot drink treatment arm only. Participants who will answer the question, 'Compared to when you had no adhesive at the start of the study day, how stable and secure does your upper denture feel?' will be evaluated for this outcome measure and will be scored on 0-4 scale as follows: 0- Much less; 1-Less; 2-Neither more or less; 3-More; 4-Much more where higher score indicates participant's perception of good denture stability.
Number of Participants who Feel Less Worried About Denture Slipping/Wobbling After Using Adhesive | Baseline, 9 hr after the BF measurement
  Denture stability and retention questionnaire will be completed by participants post dinner and hot drink after 9hr BF measurement for investigational adhesive + hot drink treatment arm only. Participants who will answer the question, 'Compared to when you had no adhesive at the start of the study day, how worried are you about your denture slipping and/or wobbling?' will be evaluated for this outcome measure and will be scored on 0-4 scale as follows: 0-Not at all worried; 1-Slightly worried; 2-Moderately worried; 3-Very worried; 4-Extremely worried, where lower score indicates participant's perception of good denture stability and retention.
Number of Participants who Feel More Confident About Having Hot Food and Drinks After Using Adhesive | Baseline, 9 hr after the BF measurement
  Denture stability and retention questionnaire will be completed by participants post dinner and hot drink after 9hr BF measurement for investigational adhesive + hot drink treatment arm only. Participants who will answer the question, 'When using this adhesive, how confident do you feel about having hot foods and drinks?' will be evaluated for this outcome measure and will be scored on 0-4 scale as follows: 0-Not at all confident; 1-Not very confident; 2-Somewhat confident; 3-Very confident; 4-Extremely confident, where higher score indicates participant's perception of good denture stability and retention.
Number of Participants who Experience Denture Adhesive OOZE After Using Adhesive | Baseline, at 0.5 hr prior to BF measurement
  Denture Adhesive Ooze Questionnaire will be completed by the participants immediately prior to the 0.5hr BF measurement for all treatment arms except the no adhesive arm. Participants who will answer the question, 'Did you experience any denture adhesive OOZE, and if so, how long after inserting your upper denture did this happen?' will be evaluated for this outcome measure and will be scored on 0-4 scale as follows: 0- Immediately; 1- Less than 10 minutes; 2- 10 to 20 minutes; 3- 20 to 30 minutes; 4- No ooze experienced, where higher score indicates participants did not experience excess adhesive ooze underneath the denture and it is well-fit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.